CLINICAL TRIAL: NCT00735007
Title: International, Multicenter, Single-arm, Open-label, 12-week Phase IIIb Study to Evaluate RebiSmart™ Suitability for Self Injection of Rebif® New Formulation (RNF) in Multidose Cartridges in Patients With Relapsing Form of Multiple Sclerosis (RMS)
Brief Title: 12-week Study to Evaluate RebiSmart™ Suitability for Self Injection in Relapsing Multiple Sclerosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28733
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rebif® New Formulation (RNF) using RebiSmartTM

INTERVENTIONS:
Drug: Rebif® New Formulation (RNF) using RebiSmartTM — RNF 44 mg, 3 times a week by subcutaneous injection.

SUMMARY:
The Electronic Device - The RebiSmart™ is an electronic injection device that is being studied for the delivery of Merck Serono's Rebif® New Formulation. The RebiSmart™ device is a stand-alone hand-held device with internal power supply. It is used for subcutaneous (under the skin) injections with single-use sterile disposable needles. The device will be kept in a storage box and placed in the refrigerator after each use.

The key features of the RebiSmart™ are as follows:

* Battery powered electromechanical automatic injector;
* Automatic needle attachment and detachment;
* Hidden needle before and after injection;
* Injection can only be initiated by pressing the injection button when in contact with the skin;
* Automatic needle insertion and injection of the preset dose into the subcutaneous (under the skin) tissue;
* Adjustable injection comfort parameters: Injection depth, needle insertion speed, medication injection speed and time that the needle remains in the skin ;
* Cartridges with 3 doses of Rebif® New Formulation; and
* Several other electronic functions including history (date and time) of cartridge changes and injections.

The Study Drug - Rebif® New Formulation (RNF) Rebif® is a medicine that is part of a family of proteins called interferon beta-1a (IFN-β-1a) molecules that play an important role in the immune system and help limit the damage that occurs with multiple sclerosis (MS). The interferon in Rebif® is like your body's own natural human interferon, but is made outside the body by a process called "recombinant DNA technology". Merck Serono International S.A. (the maker of Rebif®) has recently updated the method to make Rebif®, and it is referred to as Rebif® New Formulation (RNF).

For the purpose of this study, the form of Rebif® New Formulation (RNF) will differ slightly from the one you currently receive. RNF will be supplied in pre-filled cartridges containing three doses of 44mcg / 0.5 ml IFN-β-1a. This is the amount required for you to administer during the course of one full week of treatment. The dosage of RNF 44mcg is injected under the skin three times per week. The RebiSmart™ device will be provided for the administration of RNF. RNF should be administered, if possible, at the same time (preferably in the late afternoon or evening) on the same three days (e.g. Monday, Wednesday, and Friday), with at least 48 hours break between each administration. You will be asked to record the time and date of each injection in the diary cards provided. You will be taught how to properly use the device to inject the medication. You will also be reminded to rotate injection sites and advised on the importance of avoiding already inflamed areas for future injections.

The goals of this research trial are:

* To evaluate if the electronic device can be used (if it is suitable) by MS patients performing self-injections of Rebif® New Formulation.
* To determine MS patients overall satisfaction of the new RebiSmart™ device by determining their ease in using it, how often side effects happen (flu-like symptoms, injection site reactions and any other overall injection issues) that they may experience while on the trial. This will be done by completion of the Patient User Trial Questionnaire and the Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ).
* To evaluate specific features of the RebiSmart™ device from the answers MS patients provide in the User Trial Questionnaire. The MS patient and the person who will trains them on the proper use of the device will complete this questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age, inclusive
* Female subjects must be neither pregnant nor breast-feeding and must lack child-bearing potential, as defined by either:

  * Post-menopausal or surgically sterile, or
  * Using a highly effective method of contraception for the duration of the study. This is defined as a method that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, and includes for instance implants, injectables, combined oral contraceptives, intra-uterine device (IUD)s, sexual abstinence or vasectomised partner.
* Have RMS according to the revised McDonald Criteria 2005
* Have disease duration for at least 3 months
* Are currently receiving RNF 44 mcg sc by Rebiject IITM (RII) tiw and have been consistently on therapy for a minimum of 6 weeks prior to Screening

Exclusion Criteria:

* Have any disease other than MS that could better explain his/her signs and symptoms
* Receive any other injectable medications on a regular basis during the week prior to the screening period or throughout the duration of the study. The administration of a single injection for treatment or prophylaxis of a condition unrelated to the patient's MS or the patient's RNF therapy (e.g., influenza or pneumococcus vaccination) will be acceptable
* Receive any MS therapy other than Rebif / RNF (e.g., other disease-modifying drug [DMD]s: immunomodulatory , immunosuppressive agents or combination therapy) within 12 months prior to study enrolment or at any time during the study
* Receive oral or systemic corticosteroids or adrenocorticotrophic hormone (ACTH) within 30 days prior to SD1
* Have inadequate liver function, defined by a alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN), or alkaline phosphatase > 2 x ULN, or total bilirubin > 2 x ULN if associated with any elevation of ALT or alkaline phosphatase
* Have inadequate bone marrow reserve, defined as a white blood cell count less than 0.5 x lower limit of normal
* Have moderate to severe renal impairment
* History of any chronic pain syndrome
* Any visual or physical impairment that precludes the subject self-injecting the treatment using the RebiSmartä

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Verdun di Cantogno, MD, Study Director — Merck Serono International, S.A., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (6):
- US Local Medical Information, Rockland, Massachusetts, United States
- Canada, Local Medical Information, Ontario, British Columbia, Quebec, Canada
- Germany, Local Medical Information, Hamburg, Ulm, Berlin, Erbach, Germany
- Italy, Local Medical Information, Chieti & Roma, Italy, Italy
- Spain, Local Medical Information, Barcelona & Madrid, Spain, Spain
- Sweden, Local Medical Information, Sweden, Sweden

REFERENCES:
- [Derived] Devonshire V, Arbizu T, Borre B, Lang M, Lugaresi A, Singer B, Verdun di Cantogno E, Cornelisse P. Patient-rated suitability of a novel electronic device for self-injection of subcutaneous interferon beta-1a in relapsing multiple sclerosis: an international, single-arm, multicentre, Phase IIIb study. BMC Neurol. 2010 Apr 30;10:28. doi: 10.1186/1471-2377-10-28. PMID 20433746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit : 30 July 2008 Last Patient Last Visit: 27 January 2009
  15 specialist neurology centres in 6 countries: Canada (3 sites), Germany(4 sites) , Italy (2 sites) , Spain(3 sites), Sweden (1 sites), USA(2 sites)
Groups:
- RebiSmart for Self-injection: Rebif New Formulation 44 mg, 3 times a week by subcutaneous injection.
Period: Overall Study
Arm/Group | RebiSmart for Self-injection
Started | 106
Completed | 101
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 21
  Canada | 16
  Spain | 24
  Germany | 26
  Italy | 14
  Sweden | 5
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 75.5 (10.1)
Heart rate [Mean (Standard Deviation); unit: beats/min] | 74.9 (9.0)
Temperature [Mean (Standard Deviation); unit: °C] | 36.40 (0.43)
Thyroid Peroxidase antibody [Mean (Standard Deviation); unit: IU/ml] | 220 (181.9)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118.4 (13.1)
Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Flu Like Symptom (FLS) Score items 13-16 [Mean (Standard Deviation); unit: units on a scale] — Intention to treat population. MSTCQ FLS Score items 13-16 has a best possible score of 4 and a worst possible score of 20.
  units on a scale | 9.5 (3.7)
Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Global Side Effects Score items 21-23 [Mean (Standard Deviation); unit: units on a scale] — Intention to treat population. MSTCQ Global Side Effects Score items 21-23 has a best possible score of 15 and a worst possible score of 3.
  units on a scale | 4.8 (1.7)
Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Site Reaction Score items 17-20 [Mean (Standard Deviation); unit: units on a scale] — Intention to treat population. MSTCQ Injection Site Reaction Score items 17-20 has a best possible score of 4 and a worst possible score of 20.
  units on a scale | 11.1 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Rating the Suitability of RebiSmart at the End of 12-week Treatment Period for Self-injecting Rebif® New Formulation (RNF).
Description: RebiSmart was evaluated as "very suitable or suitable"; "a little suitable"; or "not suitable at all" for self-injecting RNF. The Patient User Trial Questionnaire (UTQ) provides confidence in the ability to evaluate the suitability of the device and ease of understanding the different features of the RebiSmart during the training session and the overall subject impression of the injection administration. Subjects completed the Patient UTQ at Study Day1, Week4, and Week12. The Trainer User UTQ provides confidence in the ability to evaluate the suitability of the RebiSmart by the trainer.
Time Frame: End of 12 week treatment period
Population: 4 subjects with missing values
Measure: Number; unit: participants
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 102
participants
  suitable or very suitable | 73
  a little suitable | 21
  not suitable at all | 8

2. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Flu Like Symptom (FLS) Score Items 13-16 at End Week 4
Description: Intention to treat population. MSTCQ FLS Score items 13-16 has a best possible score of 4 and a worst possible score of 20.
Time Frame: at the end of week 4 of treatment
Population: 3 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 103
MSTCQ Score (units on a scale) | 8.8 (3.9)

3. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Flu Like Symptom (FLS) Score Items 13-16 at End Week 8
Description: as for outcome 2
Time Frame: at the end of week 8 of treatment
Population: 6 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 100
MSTCQ Score (units on a scale) | 8.8 (3.8)

4. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Flu Like Symptom (FLS) Score Items 13-16 at End Week 12
Description: as for outcome 2
Time Frame: at the end of week 12 of treatment
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 106
MSTCQ Score (units on a scale) | 9.0 (3.8)

5. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Site Reaction Score Items 17-20 at End Week 4
Description: Intention to treat population. MSTCQ InjectionSite Reaction Score items 17-20 has a best possible score of 4 and a worst possible score of 20.
Time Frame: at the end of week 4 of treatment
Population: 3 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 103
MSTCQ Score (units on a scale) | 11.4 (3.2)

6. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Site Reaction Score Items 17-20 at End Week 8
Description: as for outcome 5
Time Frame: at the end of week 8 of treatment
Population: 6 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 100
MSTCQ Score (units on a scale) | 11.3 (3.5)

7. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Site Reaction Score Items 17-20 at End Week 12
Description: as for outcome 5
Time Frame: at the end of week 12 of treatment
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 106
MSTCQ Score (units on a scale) | 11.4 (3.4)

8. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Global Side Effects Score Items 21-23 at End Week 4
Description: Intention to treat population. MSTCQ Global Side Effects Score items 21-23 has a best possible score of 15 and a worst possible score of 3.
Time Frame: at the end of week 4 of treatment
Population: 3 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 103
MSTCQ Score (units on a scale) | 5.5 (2.4)

9. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Global Side Effects Score Items 21-23 at End Week 8
Description: as for outcome 8
Time Frame: at the end of week 8 of treatment
Population: 6 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 100
MSTCQ Score (units on a scale) | 5.2 (2.2)

10. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Global Side Effects Score Items 21-23 at End Week 12
Description: as for outcome 8
Time Frame: at the end of week 12 of treatment
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 106
MSTCQ Score (units on a scale) | 5.6 (2.6)

11. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Issues Score Item 34 at End Week 4
Description: Intention to treat population. MSTCQ Injection Issues Score item 34: +5 is the best possible score (much better), -5 is the worst possible score (much worse), zero is neutral (no change)
Time Frame: at the end of week 4 of treatment
Population: 3 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 103
MSTCQ Score (units on a scale) | 0.2 (2.5)

12. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Issues Score Item 34 at End Week 8
Description: as for outcome 11
Time Frame: at the end of week 8 of treatment
Population: 5 subjects with missing values
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 101
MSTCQ Score (units on a scale) | 0.1 (1.9)

13. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Injection Issues Score Item 34 at End Week 12
Description: as for outcome 11
Time Frame: at the end of week 12 of treatment
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: MSTCQ Score (units on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 106
MSTCQ Score (units on a scale) | 0.2 (2.0)

14. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Benefit Item 35 at End Week 4
Description: Intention to treat population. MSTCQ Injection Issues Score item 35 - Most important benefit of the RebiSmart injection system: Fewer injection site reactions; less injection pain; fewer flu-like symptoms; fewer physical side effects; or overall convenience.
Time Frame: at the end of week 4 of treatment
Population: 21 subjects with missing values
Measure: Number; unit: participants
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 85
participants
  fewer injection site reactions | 13
  less injection pain | 17
  fewer flu-like symptoms | 9
  fewer physical side effects | 5
  overall convenience | 50

15. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Benefit Item 35 at End Week 8
Description: as for outcome 14
Time Frame: at the end of week 8 of treatment
Population: 21 subjects with missing values
Measure: Number; unit: participants
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 85
participants
  fewer injection site reactions | 8
  less injection pain | 13
  fewer flu-like symptoms | 6
  fewer physical side effects | 8
  overall convenience | 59

16. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Benefit Item 35 at End Week 12
Description: as for outcome 14
Time Frame: at the end of week 12 of treatment
Population: 21 subjects with missing values
Measure: Number; unit: participants
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 85
participants
  fewer injection site reactions | 6
  less injection pain | 11
  fewer flu-like symptoms | 6
  fewer physical side effects | 5
  overall convenience | 63

17. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Pain Rating Scale Item 37 at End Week 4
Description: Intention to treat population. MSTCQ Pain Rating Scale item 37. Visual Analogue Scale 0mm (No pain) to 100mm (Worst possible pain)
Time Frame: at the end of week 4 of treatment
Population: 4 subjects with missing values
Measure: Mean (Standard Deviation); unit: mm (on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 102
mm (on a scale) | 30.2 (24.6)

18. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Pain Rating Scale Item 37 at End Week 8
Description: as for outcome 17
Time Frame: at the end of week 8 of treatment
Population: 5 subjects with missing values
Measure: Mean (Standard Deviation); unit: mm (on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 101
mm (on a scale) | 30.8 (24.9)

19. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Pain Rating Scale Item 37 at End Week 12
Description: as for outcome 17
Time Frame: at the end of week 12 of treatment
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: mm (on a scale)
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 106
mm (on a scale) | 30.0 (25.1)

20. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Pain Rating Grade Item 38 at End Week 4
Description: Intention to treat population. MSTCQ Pain Rating Grade item 38. Rated as No pain; Mild; Discomforting; Distressing; or Horrible Excruciating
Time Frame: at the end of week 4 of treatment
Population: 5 subjects with missing values
Measure: Number; unit: participants
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 101
participants
  No pain | 18
  Mild | 44
  Discomforting | 26
  Distressing | 11
  Horrible Excruciating | 2

21. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Pain Rating Grade Item 38 at End Week 8
Description: as for outcome 20
Time Frame: at the end of week 8 of treatment
Population: 5 subjects with missing values
Measure: Number; unit: participants
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 101
participants
  No pain | 17
  Mild | 46
  Discomforting | 25
  Distressing | 12
  Horrible Excruciating | 1

22. Secondary Outcome: Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Pain Rating Grade Item 38 at End Week 12
Description: as for outcome 20
Time Frame: at the end of week 12 of treatment
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | RebiSmart for Self-injection
Number analyzed (Participants) | 106
participants
  No pain | 18
  Mild | 42
  Discomforting | 31
  Distressing | 11
  Horrible Excruciating | 4

23. Secondary Outcome: The Incidence of Predefined Injection Site Reactions, MSTCQ Scores, Side Effects, McGill Pain Questionnaire, Visual Analog Scale, and Rating of Pain Regarding Injection Pain Following RNF Administration With RebiSmart at 12-week Treatment Period.
Description: Information on these outcomes is shown separately above, apart from information on the incidence of injection site related adverse events which is shown in the Adverse Events section
Time Frame: at the end of weeks 4, 8, and 12 of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The timeframe over which adverse events were collected was during the 12-week treatment period.
Description: Intent to treat population. The Other Adverse Events table shows all adverse events occuring a frequency equal to or greater than the reporting threshold.
Arm/Group | RebiSmart for Self-injection
Serious Adverse Events (participants affected / at risk) | 6/106
Other Adverse Events (participants affected / at risk) | 67/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RebiSmart for Self-injection (N=106)
Adverse drug reaction (General disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Breast infection (Infections and infestations) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Myocardial disorders (Cardiac disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RebiSmart for Self-injection (N=106)
Adverse drug reaction (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Borrelia infection (Infections and infestations) | 1 (1)
Breast infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3)
Chills (General disorders) | 3 (7)
Facial palsy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 12 (25)
Impaired healing (General disorders) | 1 (1)
Influenza (Infections and infestations) | 4 (4)
Infuenza like illness (General disorders) | 22 (54)
Injection site erythema (General disorders) | 2 (2)
Injection site extravasation (General disorders) | 1 (1)
Injection site irritation (General disorders) | 2 (2)
Injection site pain (General disorders) | 3 (3)
Monoparesis (Nervous system disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Nasopharyngitis (Infections and infestations) | 10 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (6)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less